CLINICAL TRIAL: NCT03068039
Title: Gastrointestinal Responses to Millet and Oats Breakfast Interventions Assessed by MRI
Brief Title: Millets and Oats MRI
Acronym: MOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: F12072016
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: MRI; blood glucose; porridge; breakfast; satiety; plasma peptides

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blind (Investigator blind)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OATS PORRIDGE (Active Comparator): Oats breakfast porridge 220 kcal served with 240 mL water
  Interventions: Other: Oats breakfast porridge
- PEARL (BAJRA) MILLET PORRIDGE (Active Comparator): Pearl (bajra) millet breakfast porridge isoenergetic (220 kcal) served with 300 mL water to make it also isovolumteric with the Oats arm
  Interventions: Other: Pearl (bajra) breakfast porridge

INTERVENTIONS:
Other: Oats breakfast porridge — Isoenergetic and isovolumteric oats breakfast porridge
  Arms: OATS PORRIDGE
Other: Pearl (bajra) breakfast porridge — Isoenergetic and isovolumteric pearl (bajra) breakfast porridge
  Arms: PEARL (BAJRA) MILLET PORRIDGE

SUMMARY:
Breakfast porridges made from milled grains are commonly eaten worldwide. Traditionally different grains are used in different countries. For example, oats are more common in the Anglo-Saxon countries whilst millet is very common in parts of India and Africa. However the nutritional value of different grains and their potential effects on the body may vary dramatically: for example the effect on blood sugar, on how fast the stomach empties after eating and how full people may feel.

RESEARCH QUESTION: The investigators think that a pearl millet breakfast will cause a smaller rise in blood sugar compared with an oat breakfast containing the same number of calories. The investigators also think that there will be a difference in how full people feel and how fast their stomach will empty. These 2 breakfasts will be fed to each one of 26 healthy volunteers, one week apart. A safe medical imaging method (MRI) will be used to look at how quickly the breakfast empty from the stomach and how this affects the small bowel. Blood glucose levels will be measured using a finger prick test (the same as used by diabetics) and some small blood samples will be taken from a vein in the arm to measure the chemicals released by the gut after feeding gut hormones.

DETAILED DESCRIPTION:
Background: Porridge breakfasts from various grains are a staple source of energy for many populations worldwide. The grains used in the porridges differ between regions, mostly due to the crops historically grown. For example, oats are more common in the Anglo-Saxon countries whilst millet is very common in parts of India and Africa. Consumption of whole grains has been associated with a variety of health benefits ranging from lower blood glucose levels, improved insulin responses, reduced cholesterol and increased diversity of the microbiota. Of particular interest to this study are recent suggestions that different grains, and particularly millet grains, may have enhanced health benefits on glucose and insulin metabolism. This may be due to different rates of digestion and absorption, for example, because of grain specific differences in starch digestibility. This could affect gastric emptying and, in turn, post prandial glycaemia and impact on satiety. However little is known about possible differences in gastric emptying between breakfast porridges from different grains and possible relationship with glucose, insulin and appetite.

The research group in Nottingham has world-leading expertise in imaging foods in the body and gastrointestinal function using non-invasive Magnetic Resonance Imaging (MRI) techniques which are particularly well suited for this kind of investigations study.

Aims:

1. to collect data on postprandial glucose levels and hormone peptide response of isoenergetic breakfast porridges made from oats and pearl millet.
2. to collect data on their gastric emptying and satiety.
3. to compare postprandial glucose levels, gastric emptying and satiety for the treatments 4. to explore relationships between glucose levels, gastric emptying and satiety.

Experimental protocol and methods: 26 healthy volunteers will participate in this 2-way study. They will attend one morning for each study, with the studies separated by approximately a week. Before the test meal, and after that approximately every 15 min for 2 hours the level of sugar (glucose) in their blood will be measured using the finger prick method, as diabetics commonly do to monitor their blood sugars. Venous blood samples will also be collected from a cannula placed in the forearm to measure gut hormones such as Peptide YY, GIP, GLP-1 and insulin. The subjects will be scanned on a research dedicated 1.5T MRI scanner. The subjects will be scanned at baseline, immediately after the test meal and then every 30 minutes for 2 hours postprandially. At baseline and every time the subjects come out of the MRI scanner they will be asaked to rate their feelings of fullness, hunger and appetite on 100mm VAS scales. Each subject will be fed two isoenergetic breakfast meals -one on each visit: Oat and Pearl millet breakfast porridge sourced from supermarkets or food manufacturers. These will be cooked in water to avoid confounding factor with milk. The test breakfast will have 220 kcal (slightly higher than a commonly recommended average portion of ~185 kcal). After this the subjects will be asked to eat as much of a pasta meal as they wish and note how much they have eaten as an objective measure of food consumption. The subjects will also complete a food diary for the rest of the day.

Measurable endpoints/ statistical power Primary endpoint: Incremental Area Under the Curve of post prandial blood glucose up to 2h (AUC2h) Secondary endpoints: Area Under the Curve of post prandial gastric volumes up to 2h (AUC2h), postprandial hormone peptide response, insulin and post prandial VAS scores up to 2h.

Descriptive and exploratory measurements: Time to Peak of blood glucose; Area Under the Curve for appetite (Fullness, Hunger, Prospective food consumption) up to 2h. The amount of pasta meal eaten ad libitum. Energy intake for the day from food diaries.

Correlations between blood, MRI and satiety data. Using Satiety data (Hunger) from our pilot study, we can calculate sample size needed using a crossover, paired design with alpha=0.05 and a power of 80% using n=26 participants.

The data will be assessed for normality using the Shapiro-Wilk test and other such methods as appropriate. Where normally distributed, endpoints will be assessed using parametric methods.

T test (primary endpoint) and AUC2h (secondary endpoints). T test of Time to Peak. Correlation (Pearson's or Spearman) between blood glucose, MRI and satiety data.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Body mass index (BMI) ≥ 18.5 and ≤ 24.9 kg/m2
* Able to give informed consent
* Apparently healthy: no medical conditions which might affect study measurements (judged by the investigators)

Exclusion Criteria:

* Restrained eating behaviour as determined by Eating habits and SCOFF screening questionnaires
* Not used to eating breakfast
* Not used to eating three meals a day
* Use of medication which interferes with study measurements (as judged by the study physician).
* Participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study.
* Reported participation in night shift work during the two weeks prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM.
* Strenuous exercise for more than10 hours per week.
* Consumption of ≥21 alcoholic drinks in a typical week
* Reported weight loss or gain ≥ 10 % of bodyweight during the six months period before the pre-study examination.
* Following a medically- or self-prescribed diet during the two weeks prior to the pre-study examination and until the end of the study
* Dislike of the products served as the dietary test treatments
* Any allergy or food intolerance to the test treatments
* Not suitable for MRI scanning (e.g., presence of metal implants, infusion pumps and pacemakers) as assessed by standard MRI safety questionnaire.
* Pregnancy declared by candidate
* Antibiotic or prescribed probiotic treatment in the past 12 weeks
* Inability to lie flat
* Not willing to eat a pasta meal
* Exceeding the scanner bed weight limit of 120kg
* Poor understanding of the spoken and/or written English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | From baseline up to 2 hours postprandially
  Incremental Area Under the Curve of post prandial blood glucose up to 2h (AUC2h) measured using finger prick method.

SECONDARY OUTCOMES:
Gastric volumes | From baseline up to 2 hours postprandially
  Area Under the Curve of post prandial gastric volumes up to 2h (AUC2h).
Hormone peptide response and insulin | From baseline up to 2 hours postprandially
  Area Under the Curve of post prandial hormone peptide response and insulin
appetite ratings VAS scores | From baseline up to 2 hours postprandially
  Area Under the Curve for appetite (Fullness, Hunger, Prospective food consumption) up to 2h.

OTHER OUTCOMES:
Time to Peak of blood glucose | Between baseline up to 2 hours postprandially
  Time to peak of post prandial blood glucose, measured using finger prick method
Ad libitum | From 12:00 hours to 13:00 hours on the study day
  The amount of pasta meal eaten ad libitum
Small bowel water content | From baseline up to 2 hours postprandially
  Area Under the Curve of post prandial small bowel water content
Motion of the stomach contents from tagged MRI images | From baseline up to 2 hours postprandially
  Motion index from standard deviation of signal intensity variation in the images
Correlations between blood, MRI and satiety data. | From baseline up to 2 hours postprandially
  Exploratory correlations between blood, MRI and satiety data

CONTACTS AND LOCATIONS:
Overall Officials: Jaber Alyami, MRes, Study Director — Nottingham Digestive Disases Centre , University of Nottingham, Nottinghamshire, United Kingdom, NG7 2UH; Luca Marciani, Principal Investigator — Nottingham Digestive Disases Centre , University of Nottingham, Nottinghamshire, United Kingdom, NG7 2UH; Moira Taylor, Principal Investigator — School of Life Sciences, University of Nottingham, Nottinghamshire, United Kingdom, NG7 2UH; Penny A Gowland, Principal Investigator — Sir Peter Mansfield Imaging Centre, University of Nottingham, Nottingham NG7 2RD, U.K.
Locations (1):
- Nottingham Digestive Disases Centre , University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Derived] Alyami J, Whitehouse E, Yakubov GE, Pritchard SE, Hoad CL, Blackshaw E, Heissam K, Cordon SM, Bligh HFJ, Spiller RC, Macdonald IA, Aithal GP, Gowland PA, Taylor MA, Marciani L. Glycaemic, gastrointestinal, hormonal and appetitive responses to pearl millet or oats porridge breakfasts: a randomised, crossover trial in healthy humans. Br J Nutr. 2019 Nov 28;122(10):1142-1154. doi: 10.1017/S0007114519001880. PMID 31709970